CLINICAL TRIAL: NCT05950646
Title: Effect of Mini-dose Dexmedetomidine-Esketamine Infusion on Sleep Quality in Older Patients Undergoing Knee or Hip Replacement Surgery: A Multicenter Randomized Controlled Trial
Brief Title: Mini-dose Dexmedetomidine-Esketamine Infusion and Perioperative Sleep Quality
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023-239
Record Dates: First submitted 2023-07-11; First posted 2023-07-18 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Old Age; Knee Replacement Surgery; Hip Replacement Surgery; Dexmedetomidine; Esketamine; Sleep Quality
Keywords: Old Age; Knee Replacement Surgery; Hip Replacement Surgery; Dexmedetomidine; Esketamine; Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Dexmedetomidine; Esketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine-esketamine combination (Experimental): Dexmedetomidine-esketamine combination will be infused at a rate of 0.01 ml/kg/h (dexmedetomidine 0.02 μg/kg/h and esketamine 5 μg/kg/h) from 8 pm in the night before surgery until 8 am in the third morning after surgery.
  Interventions: Drug: Dexmedetomidine; Drug: Esketamine
- Normal saline (Placebo Comparator): Placebo (normal saline) will be infused at a rate of 0.01 ml/kg/h from 8 pm in the night before surgery until 8 am in the third morning after surgery.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine will be infused at a rate of 0.01 ml/ kg/h (0.02 μg/kg/h) from 8 pm in the night before surgery until 8 am in the third morning after surgery.
  Arms: Dexmedetomidine-esketamine combination
Drug: Esketamine — Esketamine will be infused at a rate of 0.01 ml/ kg/h (5 μg/kg/h) from 8 pm in the night before surgery until 8 am in the third morning after surgery.
  Arms: Dexmedetomidine-esketamine combination
Drug: Normal saline — Normal saline will be infused at a rate of 0.01 ml/ kg/h from 8 pm in the night before surgery until 8 am in the third morning after surgery.
  Arms: Normal saline

SUMMARY:
Sleep disturbances are prevalent in older patients with osteoarthrosis or fracture who are scheduled for knee or hip replacement surgery. The occurrence of sleep disturbances is associated with worse outcomes including increased risk of delirium and cardiac events, and worsened functional recovery. Dexmedetomidine is a highly selective α2-adrenergic agonist with sedative, anxiolytic, and analgesic properties. It exerts sedative effects via activating the endogenous sleep pathways and produces a state like non-rapid eye movement sleep, which is different from opioid- and benzodiazepine-induced sedation. Esketamine is a N-methyl-D-aspartic acid receptor antagonist and has been used as an anesthetic and analgesic. Recent studies showed that low-dose esketamine has anti-depressive and sleep-promoting effects. The investigators suppose that mini-dose dexmedetomidine-esketamine combined infusion at night can improve perioperative sleep quality in patients scheduled for knee or hip replacement surgery.

DETAILED DESCRIPTION:
Sleep is a naturally recurring state characterized by lowered consciousness, reduced sensory and voluntary activity, and inhibited interaction with surroundings. Normal sleep has a particular structure and a significant circadian rhythm, and is vital for both physical and mental health. Evidence shows that the restorative effect of sleep may be a consequence of the enhanced removal of potentially neurotoxic waste products like β-amyloid or tau protein via the glymphatic system in the neurological system.

Sleep disturbances frequently occur in elderly patients with chronic pain and complicated comorbidity. A meta-analysis shows that in adults, total sleep time, sleep efficiency, percentage of slow-wave sleep, and percentage of rapid eye movement (REM) sleep significantly decrease, while sleep latency, percentage of stage 1 non-REM sleep, percentage of stage 2 non-REM sleep, and wake after sleep onset significantly increase with ageing. Coexisting disease such as asthma and obstructive sleep apnea are also associated with poorer sleep quality, as manifested by increased stage 1 and 2 non-REM sleep, and decreased REM sleep. Furthermore, pain and sleep disturbances are closely correlated, and sleep disturbances frequently accompany pain from osteoarthritis (OA) or fracture in elderly patients who are scheduled for knee or hip arthroplasty.

Sleep disturbances are common after major surgery owing to preoperative comorbidity, residual anesthetic effects, surgical trauma, postoperative pain, use of analgesics, and hospital environment. Patients may report shortened total sleep time, increased number of arousals/awakenings, lowered subjective sleep quality, and sometimes nightmares. Polysomnographic monitoring reveals sleep deprivation, sleep fragmentation, altered sleep architecture (increased light sleep, decreased or disappeared deep and rapid eye movement sleep), and disordered circadian rhythm. Considering the importance of normal sleep for human health, it is not surprising that sleep disturbances may produce harmful effects on patients' recovery. Indeed, emerging evidence suggests that sleep disturbances are associated with increased sensitivity to pain, higher inflammation, more delirium, more cardiovascular events, and prolonged hospital stay.

Dexmedetomidine, an α2 adrenoceptor agonist with both sedative and analgesic properties, has increasingly been used. Unlike other sedative agents, dexmedetomidine exerts its sedative effects through an endogenous sleep-promoting pathway and preserves sleep architecture to some degree. In a recent study of mechanically ventilated ICU patients, nighttime infusion of a sedative dose of dexmedetomidine (median infusion rate 0.6 μg/kg/h [interquartile range, 0.4 to 0.7]) helped preserve the circadian of sleep and improved the sleep architecture by increasing sleep efficiency and stage 2 non-REM sleep. In our previous study of non-mechanically ventilated ICU patients, nighttime infusion of low-dose of dexmedetomidine (0.1 μg/kg/h) improved the sleep architecture by increasing sleep efficiency and stage 2 non-REM sleep. Our subsequent large randomized controlled trial showed that low-dose night-time infusion of dexmedetomidine improved sleep and decreased the incidence of delirium.

Esketamine is a N-methyl-D-aspartic acid receptor antagonist and has been used as an anesthetic and analgesic. Recent studies showed that low-dose esketamine has anti-depressive and sleep-promoting effects.

We suppose that, for older patients with osteoarthrosis or fracture who are scheduled for knee or hip replacement surgery, nighttime infusion of mini-dose dexmedetomidine-esketamine combination starting from the preoperative night and continuing in the postoperative period may improve sleep quality and postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years and <90 years;
* Scheduled to undergo unilateral knee or hip arthroplasty.

Exclusion Criteria:

* Refuse to participate;
* Hypnotic therapy for sleep disorders within 3 months;
* Preoperative history of schizophrenia, epilepsy, Parkinson's disease, or myasthenia gravis;
* Diagnosed as obstructive sleep apnea, or at high risk of moderate to severe obstructive sleep apnea according to the Stop-Bang questionnaire;
* Inability to communicate in the preoperative period because of coma, profound dementia, or language barrier;
* Sick sinus syndrome, severe sinus bradycardia (heart rate <50 beats/min), or atrioventricular block above grade II without pacemaker implanted;
* Severe hepatic dysfunction (Child-Pugh class C), renal dysfunction (required preoperative dialysis), or expected survival ≤24 hours;
* Receiving treatment with dexmedetomidine, clonidine, or esketamine;
* Allergy to dexmedetomidine or esketamine.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Subjective sleep quality in the night of surgery. | The night on the day of surgery.
  Subjective sleep quality will be assessed in the next morning (between 8:00 am to 10:00 am) with the Richards-Campbell Sleep Questionnaire (RCSQ). The RCSQ is a self-reported measure that evaluated perception of nighttime sleep in five items, including sleep depth, sleep latency, number of awakenings, returning to sleep, and overall sleep quality. Each item was assessed with a 100-millimeter visual analog scale (score ranges from 0 to 100, with higher scores representing better sleep). The mean score of the five items represents the overall RCSQ score.

SECONDARY OUTCOMES:
Total sleep time per night during the perioperative period. | From the night before surgery until the second night after surgery.
  Objective sleep quality will be monitored with the SOMNOtouch NIBP (Somnomedics GmbH, Randersacker, Germany) from 8:00 pm to 8:00 am from the night before surgery until the fifth night after surgery. Total sleep time is defined as the sum in time scored as asleep.
Sleep efficiency per night during the perioperative period. | From the night before surgery until the second night after surgery.
  Objective sleep quality will be monitored with SOMNOtouch NIBP (Somnomedics GmbH, Randersacker, Germany) from 8:00 pm to 8:00 am from the night before surgery until the fifth night after surgery. Sleep efficiency is defined as the ratio of total sleep time/time in bed.
Sleep onset latency per night during the perioperative period. | From the night before surgery until the second night after surgery.
  Objective sleep quality will be monitored with SOMNOtouch NIBP (Somnomedics GmbH, Randersacker, Germany) from 8:00 pm to 8:00 am from the night before surgery until the fifth night after surgery. Sleep onset latency is defined as time difference between time to bed and sleep start.
Wake after sleep onset per night during the perioperative period. | From the night before surgery until the second night after surgery.
  Objective sleep quality will be monitored with SOMNOtouch NIBP (Somnomedics GmbH, Randersacker, Germany) from 8:00 pm to 8:00 am from the night before surgery until the fifth night after surgery. Wake after sleep onset is defined as the total time scored as awake between sleep start and sleep end.
Subjective sleep quality during the perioperative period. | From the night before surgery until the fifth night after surgery.
  Subjective sleep quality will be assessed daily in the next morning (between 8:00 am to 10:00 am) using the Richards-Campbell Sleep Questionnaire (RCSQ).

OTHER OUTCOMES:
Cerebrospinal fluid and blood proteomics examination (selected patients). | During anesthesia.
  Cerebrospinal fluid and blood sample will be collected. Deep proteome analysis will be performed to detect protein biomarkers including amyloid-beta, total tau, and phosphorylated tau.
Intensity of pain during the first 5 postoperative days. | Up to 5 days after surgery.
  Intensity of pain will be assessed twice after surgery with the Numeric Rating Scale (an 11- point scale where 0 indicates no pain and 10 the worst pain).
Use of supplemental analgesics | Up to 5 days after surgery.
  Include opioids and non-opioid analgesics.
The incidence of delirium within 5 days after surgery. | Up to 5 days after surgery.
  Delirium is assessed twice daily (8:00-10:00 am and 6:00-8:00 pm) with the 3-minute diagnostic interview for Confusion Assessment Method-defined delirium (3D-CAM).
Length of stay in hospital after surgery. | Up to 30 days after surgery.
  Length of stay in hospital after surgery.
Occurrence of non-delirium complications within 30 days after surgery. | Up to 30 days after surgery.
  Indicated new-onset conditions other than delirium that required therapeutic intervention within 30 days after surgery.
Subjective sleep quality (Pittsburgh Sleep Quality Index) at 3 months after surgery. | At the end of the 3rd month after surgery.
  Subjective sleep quality at 30 days after surgery will be assessed with the Pittsburgh Sleep Quality Index. This is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score.
Cognitive function at 3 months after surgery. | At the end of the 3rd month after surgery.
  Cognitive function is assessed with the modified Telephone Interview for Cognitive Status.
Health related quality of life at 3 months after surgery. | At the end of the 3rd month after surgery.
  Health related quality of life is assessed with the short-form 36-item health survey questionnaire (SF-36). The SF-36 scale measures eight aspects of health status, i.e., physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. It also measures changes of subjective healthy status during the last year (reported health transition). The scores of the above 9 items are calculated separately with scores range from 0 to 100, with higher score indicating better quality.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD,PhD, Principal Investigator — Peking University First Hospital
Locations (2):
- China (2):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel JM. Sleep viewed as a state of adaptive inactivity. Nat Rev Neurosci. 2009 Oct;10(10):747-53. doi: 10.1038/nrn2697. Epub 2009 Aug 5. PMID 19654581
- [Background] Berry RB. Fundamentals of sleep medicine. Philadelphia: Elsevier Saunders; 2012.
- [Background] Xie L, Kang H, Xu Q, Chen MJ, Liao Y, Thiyagarajan M, O'Donnell J, Christensen DJ, Nicholson C, Iliff JJ, Takano T, Deane R, Nedergaard M. Sleep drives metabolite clearance from the adult brain. Science. 2013 Oct 18;342(6156):373-7. doi: 10.1126/science.1241224. PMID 24136970
- [Background] Ratner V, Gao Y, Lee H, Elkin R, Nedergaard M, Benveniste H, Tannenbaum A. Cerebrospinal and interstitial fluid transport via the glymphatic pathway modeled by optimal mass transport. Neuroimage. 2017 May 15;152:530-537. doi: 10.1016/j.neuroimage.2017.03.021. Epub 2017 Mar 18. PMID 28323163
- [Background] Irwin MR. Sleep and inflammation: partners in sickness and in health. Nat Rev Immunol. 2019 Nov;19(11):702-715. doi: 10.1038/s41577-019-0190-z. PMID 31289370
- [Background] Ohayon MM, Carskadon MA, Guilleminault C, Vitiello MV. Meta-analysis of quantitative sleep parameters from childhood to old age in healthy individuals: developing normative sleep values across the human lifespan. Sleep. 2004 Nov 1;27(7):1255-73. doi: 10.1093/sleep/27.7.1255. PMID 15586779
- [Background] Sundbom F, Janson C, Malinovschi A, Lindberg E. Effects of Coexisting Asthma and Obstructive Sleep Apnea on Sleep Architecture, Oxygen Saturation, and Systemic Inflammation in Women. J Clin Sleep Med. 2018 Feb 15;14(2):253-259. doi: 10.5664/jcsm.6946. PMID 29394961
- [Background] Andrechuk CR, Ceolim MF. Sleep quality and adverse outcomes for patients with acute myocardial infarction. J Clin Nurs. 2016 Jan;25(1-2):223-30. doi: 10.1111/jocn.13051. PMID 26769209
- [Background] Onen SH, Onen F, Courpron P, Dubray C. How pain and analgesics disturb sleep. Clin J Pain. 2005 Sep-Oct;21(5):422-31. doi: 10.1097/01.ajp.0000129757.31856.f7. PMID 16093748
- [Background] Lintzeris N, Moodley R, Campbell G, Larance B, Bruno R, Nielsen S, Degenhardt L. Sleep Quality Among People Living With Chronic Noncancer Pain: Findings From the Pain and Opioids IN Treatment (POINT) Cohort. Clin J Pain. 2016 May;32(5):380-7. doi: 10.1097/AJP.0000000000000282. PMID 26218004
- [Background] Er MS, Altinel EC, Altinel L, Erten RA, Eroglu M. An assessment of sleep quality in patients undergoing total knee arthroplasty before and after surgery. Acta Orthop Traumatol Turc. 2014;48(1):50-4. doi: 10.3944/AOTT.2014.3163. PMID 24643100
- [Background] Sasaki E, Tsuda E, Yamamoto Y, Maeda S, Inoue R, Chiba D, Okubo N, Takahashi I, Nakaji S, Ishibashi Y. Nocturnal knee pain increases with the severity of knee osteoarthritis, disturbing patient sleep quality. Arthritis Care Res (Hoboken). 2014 Jul;66(7):1027-32. doi: 10.1002/acr.22258. PMID 24470323
- [Background] Rampes S, Ma K, Divecha YA, Alam A, Ma D. Postoperative sleep disorders and their potential impacts on surgical outcomes. J Biomed Res. 2019 Aug 29;34(4):271-280. doi: 10.7555/JBR.33.20190054. PMID 32519977
- [Background] Gogenur I, Wildschiotz G, Rosenberg J. Circadian distribution of sleep phases after major abdominal surgery. Br J Anaesth. 2008 Jan;100(1):45-9. doi: 10.1093/bja/aem340. Epub 2007 Nov 23. PMID 18037670
- [Background] Yilmaz H, Iskesen I. Follow-up with objective and subjective tests of the sleep characteristics of patients after cardiac surgery. Circ J. 2007 Oct;71(10):1506-10. doi: 10.1253/circj.71.1506. PMID 17895541
- [Background] Knill RL, Moote CA, Skinner MI, Rose EA. Anesthesia with abdominal surgery leads to intense REM sleep during the first postoperative week. Anesthesiology. 1990 Jul;73(1):52-61. doi: 10.1097/00000542-199007000-00009. PMID 2360740
- [Background] Fatah RMN, Abdulrahman BB. A sleep disturbance after total knee arthroplasty. J Family Med Prim Care. 2020 Jan 28;9(1):119-124. doi: 10.4103/jfmpc.jfmpc_595_19. eCollection 2020 Jan. PMID 32110576
- [Background] Mukartihal RK, Angadi DS, Mangukiya HJ, Singh NK, Varad S, Ramesh PA, Patil SS. Temporal changes in sleep quality and knee function following primary total knee arthroplasty: a prospective study. Int Orthop. 2022 Feb;46(2):223-230. doi: 10.1007/s00264-021-05192-1. Epub 2021 Aug 27. PMID 34453191
- [Background] Sipila RM, Kalso EA. Sleep Well and Recover Faster with Less Pain-A Narrative Review on Sleep in the Perioperative Period. J Clin Med. 2021 May 7;10(9):2000. doi: 10.3390/jcm10092000. PMID 34066965
- [Background] Bjurstrom MF, Irwin MR, Bodelsson M, Smith MT, Mattsson-Carlgren N. Preoperative sleep quality and adverse pain outcomes after total hip arthroplasty. Eur J Pain. 2021 Aug;25(7):1482-1492. doi: 10.1002/ejp.1761. Epub 2021 Mar 23. PMID 33682177
- [Background] Slatore CG, Goy ER, O'hearn DJ, Boudreau EA, O'Malley JP, Peters D, Ganzini L. Sleep quality and its association with delirium among veterans enrolled in hospice. Am J Geriatr Psychiatry. 2012 Apr;20(4):317-26. doi: 10.1097/JGP.0b013e3182487680. PMID 22367162
- [Background] Cho MR, Song SK, Ryu CH. Sleep Disturbance Strongly Related to the Development of Postoperative Delirium in Proximal Femoral Fracture Patients Aged 60 or Older. Hip Pelvis. 2020 Jun;32(2):93-98. doi: 10.5371/hp.2020.32.2.93. Epub 2020 Jun 15. PMID 32566540
- [Background] Hunt JO, Hendrata MV, Myles PS. Quality of life 12 months after coronary artery bypass graft surgery. Heart Lung. 2000 Nov-Dec;29(6):401-11. doi: 10.1067/mhl.2000.110578. PMID 11080320
- [Background] Fernandes NM, Nield LE, Popel N, Cantor WJ, Plante S, Goldman L, Prabhakar M, Manlhiot C, McCrindle BW, Miner SE. Symptoms of disturbed sleep predict major adverse cardiac events after percutaneous coronary intervention. Can J Cardiol. 2014 Jan;30(1):118-24. doi: 10.1016/j.cjca.2013.07.009. Epub 2013 Oct 16. PMID 24140074
- [Background] Keating GM. Dexmedetomidine: A Review of Its Use for Sedation in the Intensive Care Setting. Drugs. 2015 Jul;75(10):1119-30. doi: 10.1007/s40265-015-0419-5. PMID 26063213
- [Background] Alexopoulou C, Kondili E, Diamantaki E, Psarologakis C, Kokkini S, Bolaki M, Georgopoulos D. Effects of dexmedetomidine on sleep quality in critically ill patients: a pilot study. Anesthesiology. 2014 Oct;121(4):801-7. doi: 10.1097/ALN.0000000000000361. PMID 24988068
- [Background] Wu XH, Cui F, Zhang C, Meng ZT, Wang DX, Ma J, Wang GF, Zhu SN, Ma D. Low-dose Dexmedetomidine Improves Sleep Quality Pattern in Elderly Patients after Noncardiac Surgery in the Intensive Care Unit: A Pilot Randomized Controlled Trial. Anesthesiology. 2016 Nov;125(5):979-991. doi: 10.1097/ALN.0000000000001325. PMID 27571256
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] Zhang DF, Su X, Meng ZT, Li HL, Wang DX, Xue-Ying Li, Maze M, Ma D. Impact of Dexmedetomidine on Long-term Outcomes After Noncardiac Surgery in Elderly: 3-Year Follow-up of a Randomized Controlled Trial. Ann Surg. 2019 Aug;270(2):356-363. doi: 10.1097/SLA.0000000000002801. PMID 29742525
- [Background] Li HJ, Li CJ, Wei XN, Hu J, Mu DL, Wang DX. Dexmedetomidine in combination with morphine improves postoperative analgesia and sleep quality in elderly patients after open abdominal surgery: A pilot randomized control trial. PLoS One. 2018 Aug 14;13(8):e0202008. doi: 10.1371/journal.pone.0202008. eCollection 2018. PMID 30106963
- [Background] Zhang ZF, Su X, Zhao Y, Zhong CL, Mo XQ, Zhang R, Wang K, Zhu SN, Shen YE, Zhang C, Wang DX. Effect of mini-dose dexmedetomidine supplemented intravenous analgesia on sleep structure in older patients after major noncardiac surgery: A randomized trial. Sleep Med. 2023 Feb;102:9-18. doi: 10.1016/j.sleep.2022.12.006. Epub 2022 Dec 20. PMID 36587547
- [Background] Persson J, Hasselstrom J, Maurset A, Oye I, Svensson JO, Almqvist O, Scheinin H, Gustafsson LL, Almqvist O. Pharmacokinetics and non-analgesic effects of S- and R-ketamines in healthy volunteers with normal and reduced metabolic capacity. Eur J Clin Pharmacol. 2002 Feb;57(12):869-75. doi: 10.1007/s002280100353. PMID 11936706
- [Background] Wang M, Zhang B, Zhou Y, Wang C, Zheng W, Liu W, Zhan Y, Lan X, Ning Y. Sleep improvement is associated with the antidepressant efficacy of repeated-dose ketamine and serum BDNF levels: a post-hoc analysis. Pharmacol Rep. 2021 Apr;73(2):594-603. doi: 10.1007/s43440-020-00203-1. Epub 2021 Jan 2. PMID 33387333
- [Background] Duncan WC, Sarasso S, Ferrarelli F, Selter J, Riedner BA, Hejazi NS, Yuan P, Brutsche N, Manji HK, Tononi G, Zarate CA. Concomitant BDNF and sleep slow wave changes indicate ketamine-induced plasticity in major depressive disorder. Int J Neuropsychopharmacol. 2013 Mar;16(2):301-11. doi: 10.1017/S1461145712000545. Epub 2012 Jun 7. PMID 22676966
- [Background] Bunney BG, Li JZ, Walsh DM, Stein R, Vawter MP, Cartagena P, Barchas JD, Schatzberg AF, Myers RM, Watson SJ, Akil H, Bunney WE. Circadian dysregulation of clock genes: clues to rapid treatments in major depressive disorder. Mol Psychiatry. 2015 Feb;20(1):48-55. doi: 10.1038/mp.2014.138. Epub 2014 Nov 4. PMID 25349171
- [Background] Bornemann-Cimenti H, Wejbora M, Michaeli K, Edler A, Sandner-Kiesling A. The effects of minimal-dose versus low-dose S-ketamine on opioid consumption, hyperalgesia, and postoperative delirium: a triple-blinded, randomized, active- and placebo-controlled clinical trial. Minerva Anestesiol. 2016 Oct;82(10):1069-1076. Epub 2016 Jun 21. PMID 27327855
- [Background] Lee KH, Lee SJ, Park JH, Kim SH, Lee H, Oh DS, Kim YH, Park YH, Kim H, Lee SE. Analgesia for spinal anesthesia positioning in elderly patients with proximal femoral fractures: Dexmedetomidine-ketamine versus dexmedetomidine-fentanyl. Medicine (Baltimore). 2020 May;99(20):e20001. doi: 10.1097/MD.0000000000020001. PMID 32443302
- [Background] Gong L, Wang Z, Fan D. Sleep Quality Effects Recovery After Total Knee Arthroplasty (TKA)--A Randomized, Double-Blind, Controlled Study. J Arthroplasty. 2015 Nov;30(11):1897-901. doi: 10.1016/j.arth.2015.02.020. Epub 2015 Feb 24. PMID 26344094
- [Background] Shen SP, Wang YJ, Zhang Q, Qiang H, Weng XS. Improved Perioperative Sleep Quality or Quantity Reduces Pain after Total Hip or Knee Arthroplasty: A Systematic Review and Meta-Analysis. Orthop Surg. 2021 Jun;13(4):1389-1397. doi: 10.1111/os.12985. PMID 34251091
- [Background] Schwenk ES, Viscusi ER, Buvanendran A, Hurley RW, Wasan AD, Narouze S, Bhatia A, Davis FN, Hooten WM, Cohen SP. Consensus Guidelines on the Use of Intravenous Ketamine Infusions for Acute Pain Management From the American Society of Regional Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists. Reg Anesth Pain Med. 2018 Jul;43(5):456-466. doi: 10.1097/AAP.0000000000000806. PMID 29870457
- [Background] Chen LX, Ji DH, Zhang F, Li JH, Cui L, Bai CJ, Liu H, Liang Y. Richards-Campbell sleep questionnaire: psychometric properties of Chinese critically ill patients. Nurs Crit Care. 2019 Nov;24(6):362-368. doi: 10.1111/nicc.12357. Epub 2018 Jul 30. PMID 30062842